CLINICAL TRIAL: NCT00000616
Title: PREMIER: Lifestyle Interventions for Blood Pressure Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 119; U01HL060574 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-11

CONDITIONS: Heart Diseases; Hypertension
MeSH Terms: conditions — Heart Diseases; Hypertension | interventions — Diet, Sodium-Restricted; Diet, Fat-Restricted; Exercise; Diet, Reducing; Ethanol

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, fat-restricted
Behavioral: exercise
Behavioral: diet, reducing
Behavioral: alcohol drinking

SUMMARY:
To compare the effectiveness of advice versus two multicomponent lifestyle interventions to control blood pressure in participants with Stage 1 hypertension or higher than optimal blood pressure.

DETAILED DESCRIPTION:
BACKGROUND:

A large body of data has been collected over the years documenting that on the one hand, reduced sodium intake, increased physical activity, weight loss, and moderate alcohol ingestion (Comprehensive Intervention) have been associated with a modest reduction of both systolic and diastolic blood pressure in with high normal and Stage 1 hypertension. On the other hand, the Dietary Approaches to Stop Hypertension (DASH) study has shown that a diet rich in fruits, vegetables, low-fat dairy products, and decreased saturated fat, total fat, and cholesterol (DASH intervention) reduced both diastolic and systolic blood pressure in similar baseline blood pressure groups.

DESIGN NARRATIVE:

A multicenter study to determine the BP-lowering effects of two multi-component lifestyle intervention programs compared with advice only. Eight hundred and ten men and women were randomly assigned to one of three treatment arms: (A) advice only; (B) comprehensive lifestyle intervention, in which participants received an intensive behavioral intervention program to facilitate achieving current lifestyle recommendations for BP control (reduced salt intake, increased physical activity, reduced alcohol intake, and weight control or weight loss if needed); and (C) comprehensive lifestyle intervention plus the DASH diet, in which participants received a behavioral intervention program to promote the DASH dietary pattern in addition to the same lifestyle recommendations for BP control. Participants were followed for 18 months. The primary outcome variable was systolic blood pressure measured at six and 18 months after randomization. Other variables included diastolic blood pressure, dietary adherence, physical activity, and onset of hypertension over the 18 months of follow-up.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Men and women, age 25 and older who were generally healthy except for higher than optimal or mildly elevated blood pressure.

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Appel — Johns Hopkins University; Pat Elmer — Kaiser Foundation Research Institute

REFERENCES:
- [Background] Appel LJ, Champagne CM, Harsha DW, Cooper LS, Obarzanek E, Elmer PJ, Stevens VJ, Vollmer WM, Lin PH, Svetkey LP, Stedman SW, Young DR; Writing Group of the PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. JAMA. 2003 Apr 23-30;289(16):2083-93. doi: 10.1001/jama.289.16.2083. PMID 12709466
- [Background] Pickering TG. Lifestyle modification and blood pressure control: is the glass half full or half empty? JAMA. 2003 Apr 23-30;289(16):2131-2. doi: 10.1001/jama.289.16.2131. No abstract available. PMID 12709472
- [Background] Svetkey LP, Harsha DW, Vollmer WM, Stevens VJ, Obarzanek E, Elmer PJ, Lin PH, Champagne C, Simons-Morton DG, Aickin M, Proschan MA, Appel LJ. Premier: a clinical trial of comprehensive lifestyle modification for blood pressure control: rationale, design and baseline characteristics. Ann Epidemiol. 2003 Jul;13(6):462-71. doi: 10.1016/s1047-2797(03)00006-1. PMID 12875806
- [Background] McGuire HL, Svetkey LP, Harsha DW, Elmer PJ, Appel LJ, Ard JD. Comprehensive lifestyle modification and blood pressure control: a review of the PREMIER trial. J Clin Hypertens (Greenwich). 2004 Jul;6(7):383-90. doi: 10.1111/j.1524-6175.2004.03147.x. PMID 15249794
- [Background] Svetkey LP, Erlinger TP, Vollmer WM, Feldstein A, Cooper LS, Appel LJ, Ard JD, Elmer PJ, Harsha D, Stevens VJ. Effect of lifestyle modifications on blood pressure by race, sex, hypertension status, and age. J Hum Hypertens. 2005 Jan;19(1):21-31. doi: 10.1038/sj.jhh.1001770. PMID 15385946
- [Background] Young DR, Aickin M, Brantley P, Elmer PJ, Harsha DW, King AC, Stevens VJ. Physical activity, cardiorespiratory fitness, and their relationship to cardiovascular risk factors in African Americans and non-African Americans with above-optimal blood pressure. J Community Health. 2005 Apr;30(2):107-24. doi: 10.1007/s10900-004-1095-7. PMID 15810564
- [Background] Ard JD, Skinner CS, Chen C, Aickin M, Svetkey LP. Informing cancer prevention strategies for African Americans: the relationship of African American acculturation to fruit, vegetable, and fat intake. J Behav Med. 2005 Jun;28(3):239-47. doi: 10.1007/s10865-005-4660-3. PMID 16015458
- [Background] Ard JD, Durant RW, Edwards LC, Svetkey LP. Perceptions of African-American culture and implications for clinical trial design. Ethn Dis. 2005 Spring;15(2):292-9. PMID 15825976
- [Result] Elmer PJ, Obarzanek E, Vollmer WM, Simons-Morton D, Stevens VJ, Young DR, Lin PH, Champagne C, Harsha DW, Svetkey LP, Ard J, Brantley PJ, Proschan MA, Erlinger TP, Appel LJ; PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on diet, weight, physical fitness, and blood pressure control: 18-month results of a randomized trial. Ann Intern Med. 2006 Apr 4;144(7):485-95. doi: 10.7326/0003-4819-144-7-200604040-00007. PMID 16585662
- [Derived] Lim YJ, van Dam RM. Impact of comprehensive lifestyle interventions on plasma branched-chain amino acid concentrations: a randomized trial. Am J Clin Nutr. 2025 Dec;122(6):1829-1835. doi: 10.1016/j.ajcnut.2025.10.008. Epub 2025 Oct 17. PMID 41106729
- [Derived] Gradinariu V, Ard J, van Dam RM. Effects of dietary quality, physical activity and weight loss on glucose homeostasis in persons with and without prediabetes in the PREMIER trial. Diabetes Obes Metab. 2023 Sep;25(9):2714-2722. doi: 10.1111/dom.15160. Epub 2023 Jun 13. PMID 37311720
- [Derived] McClure ST, Rebholz CM, Mitchell DC, Selvin E, Appel LJ. The association of dietary phosphorus with blood pressure: results from a secondary analysis of the PREMIER trial. J Hum Hypertens. 2020 Feb;34(2):132-142. doi: 10.1038/s41371-019-0231-x. Epub 2019 Aug 21. PMID 31435005
- [Derived] Chen L, Caballero B, Mitchell DC, Loria C, Lin PH, Champagne CM, Elmer PJ, Ard JD, Batch BC, Anderson CA, Appel LJ. Reducing consumption of sugar-sweetened beverages is associated with reduced blood pressure: a prospective study among United States adults. Circulation. 2010 Jun 8;121(22):2398-406. doi: 10.1161/CIRCULATIONAHA.109.911164. Epub 2010 May 24. PMID 20497980
- [Derived] Chen L, Appel LJ, Loria C, Lin PH, Champagne CM, Elmer PJ, Ard JD, Mitchell D, Batch BC, Svetkey LP, Caballero B. Reduction in consumption of sugar-sweetened beverages is associated with weight loss: the PREMIER trial. Am J Clin Nutr. 2009 May;89(5):1299-306. doi: 10.3945/ajcn.2008.27240. Epub 2009 Apr 1. PMID 19339405
- See also: Related Info — http://www.kpchr.org/premier